CLINICAL TRIAL: NCT05626621
Title: Efficacy of Azelastine and Mometasone Irrigation in Comparison to Nasal Sprays in Patients With Chronic Rhinitis
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Endeavor Health (Other)
Responsible Party: Principal Investigator, Auddie Sweis, Principal Investigator, Endeavor Health
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EH22-362
Record Dates: First submitted 2022-11-15; First posted 2022-11-25 (Actual); Last update posted 2023-07-28 (Actual); Status verified 2023-07

CONDITIONS: Chronic Rhinitis
Keywords: mometasone; azelastine; irrigation; topical therapy; nasal spray; chronic rhinitis
MeSH Terms: interventions — azelastine; Nasal Sprays; Mometasone Furoate; Nasal Lavage

STUDY DESIGN:
Who Masked: Participant
Masking Description: Arm 1 is not blinded because this is the spray group. Arm 2 and 3 are blinded because these are both irrigation groups-either just mometasone or mometasone combined with azelastine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Azelastine and Mometasone Nasal Spray (Active Comparator): The study intervention will be saline irrigation (240 mL) followed by azelastine spray (137 mcg/spray) and mometasone spray (50 mcg/spray). Participants will have to dissolve the salt packet in a 240 mL sinus rinse bottle to create the saline solution. All participants will be instructed to perform the following twice a day: irrigation of right and left nasal cavity with half of the saline solution for each side followed by 2 sprays per nostril of both of the nasal sprays.
  Interventions: Drug: Azelastine (137 mcg/spray) Nasal Spray and Mometasone (50 mcg/spray) Nasal Spray
- Mometasone Nasal Irrigation (Experimental): The study intervention will be mometasone (1 mg/capsule). Participants will be required to dissolve the contents of the capsule into a 240 mL sinus rinse bottle along with the salt packet to create the rinse solution. All participants will be instructed to perform the following twice a day: irrigation of right and left nasal cavity with half of the rinse solution for each side.
  Interventions: Drug: Mometasone Nasal Irrigation (1 mg capsule)
- Azelastine and Mometasone Nasal Irrigation (Experimental): The study intervention will be azelastine (1mg) and mometasone (1 mg). The azelastine and mometasone will be provided in one capsule identical to the mometasone capsule. Participants will be required to dissolve the contents of the capsule into a 240 mL sinus rinse bottle along with the salt packet to create the rinse solution. All participants will be instructed to perform the following twice a day: irrigation of right and left nasal cavity with half of the rinse solution for each side.
  Interventions: Drug: Mometasone (1 mg) and Azelastine (1 mg) Nasal Irrigation

INTERVENTIONS:
Drug: Azelastine (137 mcg/spray) Nasal Spray and Mometasone (50 mcg/spray) Nasal Spray — Participants will follow this medication regimen for 6 months.
  Other Names: Astelin, Nasonex
  Arms: Azelastine and Mometasone Nasal Spray
Drug: Mometasone Nasal Irrigation (1 mg capsule) — Participants will follow this medication regimen for 6 months.
  Other Names: Nasonex
  Arms: Mometasone Nasal Irrigation
Drug: Mometasone (1 mg) and Azelastine (1 mg) Nasal Irrigation — Participants will follow this medication regimen for 6 months.
  Other Names: Astelin, Nasonex
  Arms: Azelastine and Mometasone Nasal Irrigation

SUMMARY:
The goal of this clinical trial is to determine the best combination of drugs and drug delivery routes to treat surgically naive chronic rhinitis patients. The main question it aims to answer is:

Do high volume, high pressure delivery mechanisms in nasal irrigation improve the efficacy of azelastine combined with nasal steroid mometasone as compared to the standard low pressure, low volume delivery mechanisms in nasal sprays?

Subjects will complete six months of one of three medication regimens:

1. Saline irrigation followed by azelastine spray and mometasone spray
2. Mometasone saline irrigation
3. Azelastine saline irrigation combined with mometasone saline irrigation.

DETAILED DESCRIPTION:
The purpose of this research is to determine whether patients with chronic rhinitis treated with mometasone and azelastine irrigations will show significant clinical improvement when compared to patients treated with mometasone and azelastine nasal sprays, and also compared to nasal irrigation with mometasone alone. Patients with chronic rhinitis require lifelong treatment options that are safe yet efficacious. Topical therapies, such as antihistamine sprays and steroid sprays as well as saline irrigations, are appropriate options as they offer symptom control without the side effects often seen in antibiotics. Azelastine and mometasone are FDA approved medications for the treatment of chronic rhinitis. Using these drugs in an off-label format in the form of irrigations rather than sprays is standard of care in rhinology. Prior studies suggest irrigation may be better than spray for topical mometasone, but more data is needed to establish the same for the combination of mometasone and azelastine. Eligible patients who are enrolled in the study will be randomized and will complete six months of one of three medication regimens. Subjects will come back to the office for three follow up visits at 4, 12, and 24 weeks after the treatment, where they will have a basic nasal endoscopy performed and be asked to complete a questionnaire about their nasal blockage symptoms.

ELIGIBILITY:
Inclusion Criteria:

* Adults 18 years and older seeking treatment for chronic rhinitis and willing to undergo six months of topical therapy.
* Diagnosis of Chronic Rhinitis.

Exclusion Criteria:

* The patient has diagnosis(es) other than chronic rhinitis that can account for his/her symptoms (septal deviation, nasal valve collapse, chronic sinusitis).
* Use of oral antihistamines or oral steroids, unless patient undergoes a 4 week washout period.
* Smokers (tobacco, marijuana, vaping, etc.).
* Known or suspected pregnancy, or lactation.
* Other medical conditions that the investigator believed would confound the study.
* Allergy to study drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2022-11-23 (Actual); Primary Completion 2025-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Improvement seen in the Sino-Nasal Outcome Test (SNOT)-22 score | Baseline, 1 month, 3 months, 6 months
  Sino-Nasal Outcome Test (SNOT-22) scores will be measured at baseline, 1 month, 3 months, and 6 months. Scores will be compared between three arms.
  The Sino-Nasal Outcome Test is a self-administered questionnaire that is used to assess nasal symptoms using a 0-5 point scale with 0=no problem, 1=very mild problem, 2=mild or slight problem, 3=moderate problem, 4=severe problem, 5=problem as bad as it can be. The SNOT-22 consists of 22 questions, rated from 0 to 5 for a minimum score of 0 to maximum score of 110, with higher scores indicating worse symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- Northshore University HealthSystem, Evanston, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Horak F. Effectiveness of twice daily azelastine nasal spray in patients with seasonal allergic rhinitis. Ther Clin Risk Manag. 2008 Oct;4(5):1009-22. doi: 10.2147/tcrm.s3229. PMID 19209282
- [Background] McTavish D, Sorkin EM. Azelastine. A review of its pharmacodynamic and pharmacokinetic properties, and therapeutic potential. Drugs. 1989 Nov;38(5):778-800. doi: 10.2165/00003495-198938050-00005. PMID 2574665
- [Background] Mosges R, Klimek L. Azelastine reduces mediators of inflammation in patients with nasal polyps. Allergy Asthma Proc. 1998 Nov-Dec;19(6):379-83. doi: 10.2500/108854198778612663. PMID 9876778
- [Background] Debbaneh PM, Bareiss AK, Wise SK, McCoul ED. Intranasal Azelastine and Fluticasone as Combination Therapy for Allergic Rhinitis: Systematic Review and Meta-analysis. Otolaryngol Head Neck Surg. 2019 Sep;161(3):412-418. doi: 10.1177/0194599819841883. Epub 2019 Apr 9. PMID 30961435
- [Background] Harvey R, Hannan SA, Badia L, Scadding G. Nasal saline irrigations for the symptoms of chronic rhinosinusitis. Cochrane Database Syst Rev. 2007 Jul 18;(3):CD006394. doi: 10.1002/14651858.CD006394.pub2. PMID 17636843
- [Background] Thomas WW 3rd, Harvey RJ, Rudmik L, Hwang PH, Schlosser RJ. Distribution of topical agents to the paranasal sinuses: an evidence-based review with recommendations. Int Forum Allergy Rhinol. 2013 Sep;3(9):691-703. doi: 10.1002/alr.21172. Epub 2013 May 31. PMID 23729216
- [Background] Smith KA, Rudmik L. Delivery of Topical Therapies. Adv Otorhinolaryngol. 2016;79:114-20. doi: 10.1159/000445145. Epub 2016 Jul 28. PMID 27466853
- [Background] Pynnonen MA, Mukerji SS, Kim HM, Adams ME, Terrell JE. Nasal saline for chronic sinonasal symptoms: a randomized controlled trial. Arch Otolaryngol Head Neck Surg. 2007 Nov;133(11):1115-20. doi: 10.1001/archotol.133.11.1115. PMID 18025315
- [Background] Derendorf H, Meltzer EO. Molecular and clinical pharmacology of intranasal corticosteroids: clinical and therapeutic implications. Allergy. 2008 Oct;63(10):1292-300. doi: 10.1111/j.1398-9995.2008.01750.x. PMID 18782107
- [Background] Bollinger ME, Diette GB, Chang CL, Stephenson JJ, Sajjan SG, Fan T, Allen-Ramey FC. Patient characteristics and prescription fill patterns for allergic rhinitis medications, with a focus on montelukast, in a commercially insured population. Clin Ther. 2010 Jun;32(6):1093-102. doi: 10.1016/j.clinthera.2010.06.003. PMID 20637964
- [Background] Papagiannopoulos P, Brown HJ, Kim YJ, Houser TK, Ganti A, Raad RA, Kuan EC, Losavio P, Batra PS, Tajudeen BA. Improved sinonasal symptom and endoscopy sinus scores with dose-escalated intranasal mometasone irrigation in patients with refractory chronic rhinosinusitis. Int Forum Allergy Rhinol. 2022 Jul;12(7):955-957. doi: 10.1002/alr.22940. Epub 2022 Jan 5. No abstract available. PMID 34894112
- [Background] Snidvongs K, Pratt E, Chin D, Sacks R, Earls P, Harvey RJ. Corticosteroid nasal irrigations after endoscopic sinus surgery in the management of chronic rhinosinusitis. Int Forum Allergy Rhinol. 2012 Sep-Oct;2(5):415-21. doi: 10.1002/alr.21047. Epub 2012 May 7. PMID 22566474
- [Background] Jiramongkolchai P, Patel S, Schneider JS. Use of Off-Label Nasal Steroid Irrigations in Long-Term Management of Chronic Rhinosinusitis. Ear Nose Throat J. 2021 Jun;100(5):329-334. doi: 10.1177/0145561321998521. Epub 2021 Mar 8. PMID 33683979
- [Background] Harvey RJ, Snidvongs K, Kalish LH, Oakley GM, Sacks R. Corticosteroid nasal irrigations are more effective than simple sprays in a randomized double-blinded placebo-controlled trial for chronic rhinosinusitis after sinus surgery. Int Forum Allergy Rhinol. 2018 Apr;8(4):461-470. doi: 10.1002/alr.22093. Epub 2018 Feb 2. PMID 29394004
- [Background] Rudmik L, Hoy M, Schlosser RJ, Harvey RJ, Welch KC, Lund V, Smith TL. Topical therapies in the management of chronic rhinosinusitis: an evidence-based review with recommendations. Int Forum Allergy Rhinol. 2013 Apr;3(4):281-98. doi: 10.1002/alr.21096. Epub 2012 Oct 8. PMID 23044832
- [Background] Park DY, Choi JH, Kim DK, Jung YG, Mun SJ, Min HJ, Park SK, Shin JM, Yang HC, Hong SN, Mo JH. Clinical Practice Guideline: Nasal Irrigation for Chronic Rhinosinusitis in Adults. Clin Exp Otorhinolaryngol. 2022 Feb;15(1):5-23. doi: 10.21053/ceo.2021.00654. Epub 2022 Feb 15. PMID 35158420
- [Background] Jiramongkolchai P, Peterson A, Kallogjeri D, Lee JJ, Kukuljan S, Liebendorfer A, Schneider JS, Klatt-Cromwell CN, Drescher AJ, Piccirillo JF. Randomized clinical trial to evaluate mometasone lavage vs spray for patients with chronic rhinosinusitis without nasal polyps who have not undergone sinus surgery. Int Forum Allergy Rhinol. 2020 Aug;10(8):936-943. doi: 10.1002/alr.22586. Epub 2020 May 29. PMID 32470217
- [Background] Harvey RJ, Debnath N, Srubiski A, Bleier B, Schlosser RJ. Fluid residuals and drug exposure in nasal irrigation. Otolaryngol Head Neck Surg. 2009 Dec;141(6):757-61. doi: 10.1016/j.otohns.2009.09.006. PMID 19932850